CLINICAL TRIAL: NCT05325502
Title: Caffeine and Reward Learning: Characterizing Behavioral Expression of Adenosine-Dopamine Interaction
Brief Title: Does Caffeine Facilitate Human Reward Learning Behaviors?
Acronym: ADoRe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yu-Shiuan Lin (Other)
Responsible Party: Sponsor-Investigator, Yu-Shiuan Lin, Postdoc researcher, Centre for Chronobiology
Organization: Centre for Chronobiology (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: CChronobiology
Record Dates: First submitted 2022-03-28; First posted 2022-04-13 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Caffeine
MeSH Terms: interventions — Caffeine; Mannitol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): 7 days placebo intake.
  Interventions: Dietary Supplement: mannitol
- Acute caffeine (Active Comparator): 6 days placebo followed by 1 day caffeine intake.
  Interventions: Dietary Supplement: caffeine; Dietary Supplement: mannitol
- Daily caffeine (Experimental): 7 days caffeine intake
  Interventions: Dietary Supplement: caffeine

INTERVENTIONS:
Dietary Supplement: caffeine — two doses per day: 200 mg caffeine in the morning; 100 mg caffeine in the afternoon
  Arms: Acute caffeine; Daily caffeine
Dietary Supplement: mannitol — two doses per day: 200 mg in the morning & 100 mg in the afternoon
  Arms: Acute caffeine; Placebo

SUMMARY:
"Learning from the rewards" is underlying the formulation of knowledge and habits in daily life. Caffeine is the most commonly used "psychoactive" substance that could change one's mind state by affecting the brain and nervous system. By such effects, caffeine enhances reward signals - dopamine - in human brains. In this research study, we will find out whether taking caffeine acutely or daily can enhance reward learning processes.

DETAILED DESCRIPTION:
Reward learning is associated with the formulation of habits, memories, and beliefs. Positive (receiving an unexpected reward) and negative reinforcement (eliminating an unwanted state) learning are primarily modulated by striatal dopamine D1 and D2 receptors. While caffeine, a psychostimulant regularly consumed by 80% worldwide population, is known to facilitate striatal dopamine signaling, the potential of caffeine on enhancing reward learning in humans remains unknown.

In this double-blind, randomized, crossover study, 36 young healthy non-smoking habitual caffeine consumers (daily dose 100 - 450 mg) who are aged between 18 and 40 will be examined. Each of the 36 participants (18 F, 18 M) will undergo an acute caffeine condition, a daily caffeine condition, and a daily placebo condition. Each condition consists of 7 days - 6 ambulatory days followed by 1 laboratory visit.

In the ambulatory part, participants will abstain from caffeine, nicotine, medications, and recreational drugs. Compliance to the interventions and abstinence of caffeine will be monitored by salivary caffeine concentration every day. Bedtime and sleep quality will be recorded in sleep diary. On the laboratory visit, participants will perform cognitive tasks on a 2.5h task battery, which includes a probabilistic selection task, a motor inhibition task, and a salience attribution test. We also measure their arousal and anxiety levels 1h after the second intake on the laboratory visit.

We will use Bayes factor analyses to test our confirmatory hypotheses (on the primary outcomes): 1) Caffeine enhances the accuracy of reward learning; 2) Daily intake of caffeine facilitates the negative reinforcement compared to acute its intake. On the secondary outcomes, we examine the exploratory hypotheses that caffeine enhances motor inhibition and motivational salience. Arousal and anxiety levels will be examined as a covariate which potentially contribute to the caffeine-induced changes in reward learning performance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 40
* Clinically healthy
* Non-smokers

Exclusion Criteria:

* Habitual caffeine intake < 100 mg or > 450 mg
* Pregnant or lactating women
* Women using hormonal contraceptives
* BMI < 18.5 or > 29.9
* Sleep disturbance or extreme chronotypes
* Nicotine or recreational drug users
* Depression, anxiety, psychosis, or neurologic disorders
* Severe heart or cardiovascular diseases
* Diabetes or metabolic diseases
* Under chronic medications
* Incapable to operate the tasks or comprehend the study information in German or English
* Users of the Bopomo alphates utilized as stimuli in the reward learning tasks
* Current enrolment in other clinical trials

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The accuracy (% of correct answers) in implicit learning through different probabilities of monetary reward feedback | 1-hour after the second intake on the 7th day
  Through a probabilistic selection task, participant will go through a training phase to learn the rules which options may be more likely to return monetary feedback, and the knowledge learned will be tested in a second phase where the task difficulty is increased, and no feedback is provided. The overall accuracy in the testing phases will be examined, as well as the accuracies in choosing or avoiding the highest and lowest reward-probability stimuli.

SECONDARY OUTCOMES:
The errors in motor inhibition (rates of false alarm) in a motor inhibition task | 1.5-hour after the second intake on the 7th day
  Through a reaction-inhibition task (Go/NoGo), participants will go through two phases of the task: 1) Only respond to a specific stimulus when it shows; 2) Respond to all stimuli except for the specific stimulus. The accuracy in motor inhibition will be indicated by the errors made in the no-go signals (i.e. false alarm).
Salience attribution behaviors | 1.5-hour after the second intake on the 7th day
  subjective perception towards the probabilities (0 -100%) of reward feedback from each choice in the probabilistic selection task.

OTHER OUTCOMES:
Self-report anxiety levels | 1-hour after the second intake on the 7th day
  State-Trait Anxiety Inventory for Adults (STAI-A) is used to examine the subjective anxiety levels in general as a trait (20 questions) and as a current state (20 questions). Participants will rate the levels using a Likert's scale (For trait - 0: Almost never, 1: Sometimes, 2: Often, 3: Almost always; For current state - 0: not at all, 1: Somewhat, 2: Moderately so, 3: Very much so).
Subjective sleepiness and alertness | 1-hour after the second intake on the 7th day
  Self-report one-question Karolinska Sleepiness Scale is used to rate the subjective sleepiness/alertness from 1 (very awake), 3 (awake), 5 (neither awake or tired), 7 (tired but no problem to stay awake), to 9 (very tired, big problem to stay awake, struggling with sleep), and 2, 4, 6, 8 for intermediate levels.
heart rate measurement | 1-hour after the second intake on the 7th day
  heart rates (per min)
blood pressure measurement | 1-hour after the second intake on the 7th day
  systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Shiuan Lin, PhD, Principal Investigator — Centre for Chronobiology, University Psychiatric Clinics Basel
Locations (1):
- Centre for Chronobiology, University Psychiatric Clinics Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
IPD data, including SAP, CSR, and analytic codes, will be made available on OSF or provided upon requests after the data requested are published.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Data will be made available after publishing (estimated to be July 2023).
Access Criteria: Researchers who are interested in using IPD data from ADoRe can either contact the Sponsor-Investigator (ys.lin@unibas.ch, Yu-Shiuan Lin, PhD) or access from ADoRe project on OSF (https://osf.io/wzf2y/). Please note that the data folder of this project will be only accessible after publishing.